CLINICAL TRIAL: NCT05625711
Title: A Prospective, Multicenter, Single-arm Clinical Study Was Conducted to Evaluate the Safety and Efficacy of Intravascular Interventional Surgical Instrument Control System and Related Consumables for Remote Delivery, Operation, and Withdrawal of Interventional Surgical Instruments (Guide Wire, Catheter, Stent, Balloon) During Endovascular Interventional Surgery for Lower Extremity Arteriosclerosis Occlusion
Brief Title: Clinical Study of Endovascular Interventional Surgical Instrument Control System and Related Consumables in Lower Extremity Arteriosclerosis Occlusive Lumen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Operation Robot Co., Ltd. (Industry)
Collaborators: Changhai Hospital (Other); Tianjin Medical University General Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMLY3001-02A
Record Dates: First submitted 2022-10-26; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Arterial Disease
Keywords: robot; peripheral arterial
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot assisted surgery (Experimental): The robot will assist doctors to complete lower limb artery surgery, including but not limited to the transfer and withdrawal of guide wire, catheter and stent
  Interventions: Device: The endovascular interventional surgical instrument control system

INTERVENTIONS:
Device: The endovascular interventional surgical instrument control system — The endovascular interventional surgical instrument control system is based on the analysis of the operation behavior of doctors and their assistants in the process of manual intervention. It simulates the coordinated movement of four manipulators, completes the advance and retreat of the catheter and guide wire cavity, and realizes the different actions of wire feeding along the tube, wire feeding along the wire, wire twisting coordination, wire replacement, stent release, etc.

SUMMARY:
This trial was a prospective, multicenter, single-group design. To undergo endovascular treatment of lower extremity arteriosclerosis obliterans After the subjects were selected and enrolled, the surgeons used the endovascular interventional surgical instrument control system developed by Shanghai Aopeng Medical Technology Co., Ltd. and the consumables of the endovascular interventional surgical instrument control system for the interventional hand Instrumentation (guide wire, catheter, stent, balloon) for remote delivery, manipulation, and withdrawal

DETAILED DESCRIPTION:
This study will verify the safety and effectiveness of the device in human peripheral vascular diseases, and verify 1. the degree of precision of its operation 2. the function of reducing radiation

ELIGIBILITY:
Inclusion Criteria:

* Meet all the following criteria to be included in the group.

  1. Age: 18 years old or above, regardless of gender.
  2. Suffering from arteriosclerosis obliterans of lower limbs, it has the indication of endovascular treatment.
  3. Volunteer to participate in the test and sign the informed consent form.

Exclusion Criteria:

* General criteria: If any of the following criteria is met, it cannot be included in the group.

  1. Pregnant or lactating women, or women of childbearing age with positive pregnancy test results.
  2. The target vessels were treated by arterial bypass grafting.
  3. Subjects participated in other clinical trials within 3 months before the screening period.
  4. Allergic history or contraindication of antiplatelet drugs, anticoagulants, anesthetics, contrast agents, scaffold materials and their coating drugs.
  5. Severe infection that is difficult to control.
* Vascular criteria: According to the CTA judgment of the diseased vessels, if any of the following criteria is met, they can not be included in the group.

  1. Perforation, dissection or aneurysm of the diseased vessel or the proximal vessel of the diseased vessel.
  2. The investigator believed that the vascular conditions were not suitable for the use of the test medical device.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Equipment technical success rate | immediately after operation
  After the endovascular treatment was completed by the surgeon using the experimental medical instrument, the proportion of subjects with successful equipment technology was achieved in the total enrolled subjects.
Surgical technique success rate | immediately after operation
  The proportion of subjects with successful surgical technique in the total enrolled subjects was achieved after the intravascular treatment of lower extremity arteriosclerosis occlusion with experimental medical instruments.

SECONDARY OUTCOMES:
Rutherford grading change | 4 days after surgery or discharge (depending on which comes first)
  The surgeon evaluated the subjects' symptoms of lower limb ischemia according to the Rutherford scale [13].
Total radiation exposure per operation (surgeon, subject operating table side) | The whole process from the beginning to the end of the operation was recorded.
  Determination method:
  1. The surgeon wears a radiation measuring device on his chest to record the total radiation exposure during surgery.
  2. Radiation measuring devices were placed around the umbilicus to record the total radiation exposure during surgery.
  Simulate the maximum total unguarded radiation exposure of the primary operator with full manual operation.
Satisfaction rate of equipment operation (convenience, stability) | Immediately after
  Scores of the Equipment Operation Evaluation Scale (Convenience, stability) used by surgeons who used experimental medical instruments to complete endovascular treatment of lower extremity arteriosclerosis occlusion.

OTHER OUTCOMES:
Incidence of adverse events (equipment-related, all-cause) | Intraoperative to postoperative 4 days or discharge day (depending on which comes first)
  The proportion of subjects with an adverse event (equipment-related, all-cause) among all subjects.
Incidence of device defects (software, hardware) | intraoperative.
  The proportion of subjects with device defects (software, hardware) in total subjects.

IPD SHARING:
Plan to Share IPD: No